CLINICAL TRIAL: NCT00472407
Title: Screening Eye Coordination Study Screening for Convergence Insufficiency in School-age Children
Brief Title: Screening for Convergence Insufficiency in School-age Children
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Marjean Kulp, Professor, Ohio State University
Other Study IDs: 2004H0161
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Convergence Insufficiency
Keywords: Normal
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this study was to assess the ability of common tests of eye alignment, convergence, and accommodation to identify children with convergence insufficiency in a school screening setting.

DETAILED DESCRIPTION:
The purpose of the Screening for Convergence Insufficiency in School-age Children study was to assess the ability of common tests of eye alignment, convergence, and accommodation to identify children with convergence insufficiency in a school screening setting (where it may not be feasible to do more than one test).

ELIGIBILITY:
Inclusion Criteria:

* Age 9 to 17 years
* Enrolled in participating school
* Parental permission, assent
* Ability to complete testing

Exclusion criteria: referral on vision screening for reduced distance visual acuity or significant uncorrected refractive error

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Of the 282 subjects included in the analysis, approximately 60% were female, 81.5% identified themselves as white, 11% as African American, 2.5% as other, and 5% did not report race. Two percent classified themselves as Hispanic or Latino, 76% reported not being Hispanic or Latino, and 22% did not report their ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjean Kulp, OD, MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

REFERENCES:
- [Background] Menjivar AM, Kulp MT, Mitchell GL, Toole AJ, Reuter K. Screening for convergence insufficiency in school-age children. Clin Exp Optom. 2018 Jul;101(4):578-584. doi: 10.1111/cxo.12661. Epub 2018 Mar 13. PMID 29534348